CLINICAL TRIAL: NCT05829837
Title: The Relationship Between Ambulation Capacity and Piriformis Muscle in Patients With Chronic Spinal Cord Injury: A Controlled, Clinical and Sonographic Study
Brief Title: The Relationship Between Ambulation Capacity and Piriformis Muscle in Patients With Chronic Spinal Cord Injury
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Gaziler Physical Medicine and Rehabilitation Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Yasin Demir, Physical Medicine and Rehabilitation Specialist, Gaziler Physical Medicine and Rehabilitation Education and Research Hospital
Other Study IDs: 37
Record Dates: First submitted 2023-04-13; First posted 2023-04-26 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Spinal Cord Injuries
Keywords: spinal cord injury; piriformis muscle; ultrasonographic evaluation
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Motor incomplete paraplegia patients: Participants with the age of 18 - 65, were selected for the study based on the following inclusion criteria: diagnosis of motor incomplete paraplegia at C or D level according to the spinal cord injury classification of the American Spinal Injury Association (ASIA) Impairment Scale with a neurological injury level between T2-S1.
  Interventions: Other: Ultrasonographic evaluation
- Non-ambulatory patients with complete spinal cord injury: Participants with the age of 18 - 65, were selected for the study based on the following inclusion criteria: non-ambulatory patients with diagnosis of motor complete paraplegia at A level according to the spinal cord injury classification of the American Spinal Injury Association (ASIA) Impairment Scale with a neurological injury level between T2-S1.
  Interventions: Other: Ultrasonographic evaluation

INTERVENTIONS:
Other: Ultrasonographic evaluation — Ultrasonographic evaluation for the thickness of piriformis muscle

SUMMARY:
Spinal cord injury (SCI) is a neurological condition causing paralysis, sensory abolishmentS and deficits including circulatory, respiratory, otonomic nervous systems, bowel and bladder functions. For patients with SCI, reducing disability, limitations of the impairment and regaining the walking ability are the main rehabilitation goals. There many prognostic factors effecting the recovery and ambulation capacity of patients.

The piriformis muscle (PM) is placed posterior to the hip joint, originates on the anterior surface of the sacrum and the sacrotuberous ligament and passes out of the pelvis through the greater sciatic foramen and separates the foramen into two spaces. The PM is the solely muscle coursing transversely throughout the greater sciatic notch, and it is the main landmark to all the important neurovasculer structures that pass from the pelvis to the gluteal region. PM serves as a hip abductor when the hip is flexed and as a hip external rotator when the hip is extended. It is innervated by branches of the posterior division of the ventral rami of S1, S2 and is the largest muscle among the deep, short external rotators of the hip and provides postural stability while standing and walking. PM has also a functional importance as it connects the sacroiliac joint and hip joint. For these reasons morphology of PM may have a clinical importance for SCI patients whom can walk.

Ultrasonography is radiation-free, noninvasive, available technique that can be used to measure muscle thickness in the monitoring and management of muscle changes during rehabilitation.

The aim of our study is to evaluate the relationship between the PM and the ambulation pattern of motor incomplete patients with chronic SCI. To the best of our knowledge, this is the first study evaluating PM in patients with SCI.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-65
* Diagnosis of motor incomplete paraplegia at C or D level according to the spinal cord injury classification of the American Spinal Injury Association (ASIA) Impairment Scale with a neurological injury level between T2-S1

Exclusion Criteria:

* Being under the age of 18 and over the age of 65
* Having joint contracture in the legs
* Unstable medical conditions
* Severe osteoporosis and high fracture risk
* Sacral or coccygeal grade 2 and higher pressure ulcers
* Peripheral neuropathy,
* Psychiatric disorder or cognitive problems

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 60 patients aged 18-65 years with diagnosis of paraplegia
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
piriformis muscle thickness with ultrasonographic evaluation | Through study completion, an average of one and a half months
  The thickness of piriformis muscle was measured by using a curvilinear transducer first placing in the lateral margin of the sacrum. The transducer was moved inferolaterally toward the greater trochanter until the medial end of the transducer remained at the lateral end of the sacrum. Piriformis muscle thickness was measured in the medial part of the tip of the ischium, that was parallel to the longitudinal plane at the sciatic notch with the patient's leg was abducted 45 degrees when the piriformis muscle was seen as a deep hypoechoic appearance beneath the gluteus maximus muscle.

CONTACTS AND LOCATIONS:
Overall Officials: Özlem Köroğlu, Principal Investigator — Gaziler Physical Medicine and Rehabilitation Education and Research Hospital